CLINICAL TRIAL: NCT05667285
Title: Chinese Post-marketing Clinical Study Project Protocol for Evaluate the Safety of BIOTRONIK Orsiro Sirolimus-Eluting Coronary Stent System
Brief Title: BIOFLOW-china Post-marketing Study (BIOTRONIK)
Acronym: BIOFLOW-China
Status: Terminated | Type: Observational
Why Stopped: According to the renewal registration certificate requirements issued by the NMPA, this product does not need to collect post-market safety data.
Sponsor: Biotronik (Beijing) Medical Device Ltd. (Industry)
Collaborators: Biotronik AG (Industry)
Responsible Party: Sponsor
Other Study IDs: C2022
Record Dates: First submitted 2022-12-09; First posted 2022-12-28 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: In-Stent Stenosis (Restenosis) of Coronary Artery Stent; Native Coronary Artery Stenosis
Keywords: Orsiro; BIOTRONIK; China; Coronary Stent System

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- BIOTRONIK Orsiro Sirolimus-Eluting Coronary Stent System: Subject implanted with BIOTRONIK Orsiro Sirolimus-Eluting Coronary Stent System in stent implantation operation.
  Interventions: Device: BIOTRONIK Orsiro Sirolimus-Eluting Coronary Stent System

INTERVENTIONS:
Device: BIOTRONIK Orsiro Sirolimus-Eluting Coronary Stent System — During the procedure, the investigator assesses the arterial diameter and lesion length either visually or using QCA to select the appropriate stent. The number of stents required for each lesion is determined by the investigator based on the specific circumstances. The length of the stent should cover from the proximal normal reference vessel to the distal normal reference vessel, ensuring complete coverage of the lesion.
  The number of stents required for each lesion is determined by the investigator based on the specific circumstances. If the first stent does not fully cover the lesion, a second or even more stents may be used. In such cases, the second or additional stents are selected by the investigator based on the specific circumstances, such as using Orsiro SES stents, unless clinically contraindicated or specifically required. Please refer to the stent's Instructions for Use for the procedure.
  If stent overlap occurs, the overlapping part should be at least 2mm.

SUMMARY:
This trial uses prospective, retrospective, observational, non-blinded, multi-center, single-arm, post-marketing hospital data collection and research methods.

The goal of this study is to assess the safety of BIOTRONIK Orsiro Sirolimus-Eluting Coronary Stent System in the Chinese patient population after marketing in China.

DETAILED DESCRIPTION:
This trial uses prospective, retrospective, observational, non-blinded, multi-center, single-arm, post-marketing hospital data collection and research methods. A total of 2,000 subjects will be enrolled from up to 15 research sites in China. Suitable subjects will be selected according to the inclusion and exclusion criteria, and those who meet the inclusion and exclusion criteria will accept follow-up after signing the informed consent form from the site ethics committee until 5 years after surgery. It is aimed to further assess the safety of BIOTRONIK Orsiro Sirolimus-Eluting Coronary Stent System in the Chinese patient population after marketing in China by observing the data collected in this trial.

ELIGIBILITY:
Inclusion Criteria:

* The subject should be 18 years or older when undergoing the procedure.
* The subject has signed the Informed Consent.
* The subject signed Informed Consent dated back within 12 months and was implanted with BIOTRONIK Orsiro Sirolimus-Eluting Coronary Stent System in stent implantation operation.

Exclusion Criteria:

* The subject has or had a life expectancy less then 12 month after treatment with BIOTRONIK Orsiro Sirolimus-Eluting Coronary Stent System in stent implantation operation.
* The subject has any known allergies to the following substances: aspirin, heparin/divalerythromycin, P2Y12 inhibitors (clopidogrel/prasugrel/ticagrelor), bivalirudin, rapamycin, L-605 cobalt-chromium (Co-Cr) alloy or its main elements (cobalt, chromium, tungsten and nickel), acrylic acid, fluoropolymer, silicon carbide, PLLA allergy or contraindications.
* The investigator judges that the subject has poor compliance and cannot complete the study as required, or other circumstances that are not suitable for participation in this study .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Sirolimus-eluting coronary stent system can improve the diameter of the coronary lumen. It is suitable for patients with ischemic heart disease symptoms caused by primary stenotic lesions and in-stent restenotic lesions (length ≤ 36 mm) dispersed within the native coronary arteries (reference vessel diameter of 2.25 mm to 4.0 mm).
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
Target lesion failure (TLF) at 1 years ± 60 days after surgery | 1 years ± 60 days after surgery
  Including cardiogenic death, target vessel Q-wave and non-Q-wave myocardial infarction, coronary artery bypass grafting (CABG), and clinically driven target lesion revascularization (TLR).

SECONDARY OUTCOMES:
Major adverse cardiac event (MACE) at 1, 2, 3, 4 and 5 years ± 60 days after surgery | 1, 2, 3, 4 and 5 years ± 60 days after surgery
  Including all-cause deaths, Q-wave or non-Q-wave myocardial infarction, and clinically driven target lesion revascularizition (TLR).
Target lesion failure (TLF) at 2, 3, 4 and 5 years ± 60 days after surgery | 2, 3, 4 and 5 years ± 60 days after surgery
  Including cardiogenic death, target vessel Q-wave and non-Q-wave myocardial infarction, coronary artery bypass grafting (CABG), and clinically driven target lesion revascularization (TLR).
Serious adverse device effects (SADEs) | 1, 2, 3, 4 and 5 years ± 60 days after surgery
  A serious adverse device effect (SADE) refers to any adverse device event that leads to the consequences and characteristics of serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Yang, Principal Investigator — The Fourth Affiliated Hospital of Harbin Medical University
Locations (2):
- China (2):
  - The 4th Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Zhejiang University Mingzhou Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided
The sponsor has exclusive ownership of the trial data and results. During the clinical trial process, the sponsor has the right to consult and use all the data and results obtained from the trial. Before the results of each site are published and/or reported, any single clinical trial site is not allowed to publish and/or report its results. The sponsor agrees that the principal investigator of the trial may publish the results of the clinical trial.

REFERENCES:
- [Background] Li C, Yang Y, Han Y, Song D, Xu J, Guan C, Gao R, Garcia-Garcia HM, Waksman R, Xu B; BIOFLOW VI Trial Investigators. Comparison of the Ultrathin Strut, Biodegradable Polymer Sirolimus-eluting Stent With a Durable Polymer Everolimus-eluting Stent in a Chinese Population: The Randomized BIOFLOW VI Trial. Clin Ther. 2020 Apr;42(4):649-660.e9. doi: 10.1016/j.clinthera.2020.02.014. Epub 2020 Apr 5. PMID 32268942
- [Background] Kandzari DE, Koolen JJ, Doros G, Garcia-Garcia HM, Bennett J, Roguin A, Gharib EG, Cutlip DE, Waksman R; BIOFLOW V Investigators. Ultrathin Bioresorbable-Polymer Sirolimus-Eluting Stents Versus Thin Durable-Polymer Everolimus-Eluting Stents for Coronary Revascularization: 3-Year Outcomes From the Randomized BIOFLOW V Trial. JACC Cardiovasc Interv. 2020 Jun 8;13(11):1343-1353. doi: 10.1016/j.jcin.2020.02.019. PMID 32499026
- [Background] Saito S, Toelg R, Witzenbichler B, Haude M, Masotti M, Salmeron R, Witkowski A, Uematsu M, Takahashi A, Waksman R, Slagboom T. BIOFLOW-IV, a randomised, intercontinental, multicentre study to assess the safety and effectiveness of the Orsiro sirolimus-eluting stent in the treatment of subjects with de novo coronary artery lesions: primary outcome target vessel failure at 12 months. EuroIntervention. 2019 Dec 6;15(11):e1006-e1013. doi: 10.4244/EIJ-D-18-01214. PMID 31235458
- [Background] Hamon M, Niculescu R, Deleanu D, Dorobantu M, Weissman NJ, Waksman R. Clinical and angiographic experience with a third-generation drug-eluting Orsiro stent in the treatment of single de novo coronary artery lesions (BIOFLOW-I): a prospective, first-in-man study. EuroIntervention. 2013 Jan 22;8(9):1006-11. doi: 10.4244/EIJV8I9A155. PMID 23339805
- [Background] Serruys PW, Silber S, Garg S, van Geuns RJ, Richardt G, Buszman PE, Kelbaek H, van Boven AJ, Hofma SH, Linke A, Klauss V, Wijns W, Macaya C, Garot P, DiMario C, Manoharan G, Kornowski R, Ischinger T, Bartorelli A, Ronden J, Bressers M, Gobbens P, Negoita M, van Leeuwen F, Windecker S. Comparison of zotarolimus-eluting and everolimus-eluting coronary stents. N Engl J Med. 2010 Jul 8;363(2):136-46. doi: 10.1056/NEJMoa1004130. Epub 2010 Jun 16. PMID 20554978
- [Background] Stone GW, Midei M, Newman W, Sanz M, Hermiller JB, Williams J, Farhat N, Mahaffey KW, Cutlip DE, Fitzgerald PJ, Sood P, Su X, Lansky AJ; SPIRIT III Investigators. Comparison of an everolimus-eluting stent and a paclitaxel-eluting stent in patients with coronary artery disease: a randomized trial. JAMA. 2008 Apr 23;299(16):1903-13. doi: 10.1001/jama.299.16.1903. PMID 18430909
- [Background] Serruys PW, Ruygrok P, Neuzner J, Piek JJ, Seth A, Schofer JJ, Richardt G, Wiemer M, Carrie D, Thuesen L, Boone E, Miquel-Herbert K, Daemen J. A randomised comparison of an everolimus-eluting coronary stent with a paclitaxel-eluting coronary stent:the SPIRIT II trial. EuroIntervention. 2006 Nov;2(3):286-94. PMID 19755303
- [Background] Tsuchida K, Piek JJ, Neumann FJ, van der Giessen WJ, Wiemer M, Zeiher AM, Grube E, Haase J, Thuesen L, Hamm CW, Veldhof S, Dorange C, Serruys PW. One-year results of a durable polymer everolimus-eluting stent in de novo coronary narrowings (The SPIRIT FIRST Trial). EuroIntervention. 2005 Nov;1(3):266-72. PMID 19758915
- [Background] Serruys PW, Ong AT, Piek JJ, Neumann FJ, van der Giessen WJ, Wiemer M, Zeiher A, Grube E, Haase J, Thuesen L, Hamm C, Otto-Terlouw PC. A randomized comparison of a durable polymer Everolimus-eluting stent with a bare metal coronary stent: The SPIRIT first trial. EuroIntervention. 2005 May;1(1):58-65. PMID 19758878
- [Background] Tsuji T, Tamai H, Igaki K, Kyo E, Kosuga K, Hata T, Okada M, Nakamura T, Komori H, Motohara S, Uehata H. Biodegradable Polymeric Stents. Curr Interv Cardiol Rep. 2001 Feb;3(1):10-17. PMID 11177716
- [Background] Ormiston JA, Serruys PW, Regar E, Dudek D, Thuesen L, Webster MW, Onuma Y, Garcia-Garcia HM, McGreevy R, Veldhof S. A bioabsorbable everolimus-eluting coronary stent system for patients with single de-novo coronary artery lesions (ABSORB): a prospective open-label trial. Lancet. 2008 Mar 15;371(9616):899-907. doi: 10.1016/S0140-6736(08)60415-8. PMID 18342684
- [Background] Grube E, Hauptmann KE, Buellesfeld L, Lim V, Abizaid A. Six-month results of a randomized study to evaluate safety and efficacy of a Biolimus A9 eluting stent with a biodegradable polymer coating. EuroIntervention. 2005 May;1(1):53-7. PMID 19758877
- [Background] Chevalier B, Serruys PW, Silber S, Garcia E, Suryapranata H, Hauptmann K, Wijns W, Schuler G, Fath-Ordoubadi F, Worthley S, Thuesen L, Meredith I, Bressers M, Nagai H, Paunovic D. Randomised comparison of Nobori, biolimus A9-eluting coronary stent with a Taxus(R), paclitaxel-eluting coronary stent in patients with stenosis in native coronary arteries: the Nobori 1 trial. EuroIntervention. 2007 Feb;2(4):426-34. PMID 19755281
- [Background] Carrie D, Khalife K, Citron B, Izaaz K, Hamon M, Juiliard JM, Leclercq F, Fourcade J, Lipiecki J, Sabatier R, Boulet V, Rinaldi JP, Mourali S, Fatouch M, El Mokhtar E, Aboujaoude G, Elbaz M, Grolleau R, Steg PG, Puel J; Benefit Evaluation of Direct Coronary Stenting Study Group. Comparison of direct coronary stenting with and without balloon predilatation in patients with stable angina pectoris. BET (Benefit Evaluation of Direct Coronary Stenting) Study Group. Am J Cardiol. 2001 Mar 15;87(6):693-8. doi: 10.1016/s0002-9149(00)01485-5. PMID 11249885
- [Background] Unverdorben M, Sattler K, Degenhardt R, Fries R, Abt B, Wagner E, Koehler H, Scholz M, Ibrahim H, Tews KH, Hennen B, Daemgen G, Berthold HK, Vallbracht C. Comparison of a silicon carbide coated stent versus a noncoated stent in humans: the Tenax- versus Nir-Stent Study (TENISS). J Interv Cardiol. 2003 Aug;16(4):325-33. doi: 10.1034/j.1600-6143.2003.08058.x. PMID 14562673
- [Background] Unverdorben M, Sippel B, Degenhardt R, Sattler K, Fries R, Abt B, Wagner E, Koehler H, Daemgen G, Scholz M, Ibrahim H, Tews KH, Hennen B, Berthold HK, Vallbracht C; Tenax versus Nir Stent Study. Comparison of a silicon carbide-coated stent versus a noncoated stent in human beings: the Tenax versus Nir Stent Study's long-term outcome. Am Heart J. 2003 Apr;145(4):e17. doi: 10.1067/mhj.2003.90. PMID 12679775
- [Background] Schampaert E, Moses JW, Schofer J, Schluter M, Gershlick AH, Cohen EA, Palisaitis DA, Breithardt G, Donohoe DJ, Wang H, Popma JJ, Kuntz RE, Leon MB; SIRIUS, E- and C-SIRIUS Investigators. Sirolimus-eluting stents at two years: a pooled analysis of SIRIUS, E-SIRIUS, and C-SIRIUS with emphasis on late revascularizations and stent thromboses. Am J Cardiol. 2006 Jul 1;98(1):36-41. doi: 10.1016/j.amjcard.2006.01.049. Epub 2006 May 4. PMID 16784917
- [Background] Schofer J, Schluter M, Gershlick AH, Wijns W, Garcia E, Schampaert E, Breithardt G; E-SIRIUS Investigators. Sirolimus-eluting stents for treatment of patients with long atherosclerotic lesions in small coronary arteries: double-blind, randomised controlled trial (E-SIRIUS). Lancet. 2003 Oct 4;362(9390):1093-9. doi: 10.1016/S0140-6736(03)14462-5. PMID 14550694
- [Background] Weisz G, Leon MB, Holmes DR Jr, Kereiakes DJ, Popma JJ, Teirstein PS, Cohen SA, Wang H, Cutlip DE, Moses JW. Five-year follow-up after sirolimus-eluting stent implantation results of the SIRIUS (Sirolimus-Eluting Stent in De-Novo Native Coronary Lesions) Trial. J Am Coll Cardiol. 2009 Apr 28;53(17):1488-97. doi: 10.1016/j.jacc.2009.01.050. PMID 19389558
- [Background] Urban P, Gershlick AH, Guagliumi G, Guyon P, Lotan C, Schofer J, Seth A, Sousa JE, Wijns W, Berge C, Deme M, Stoll HP; e-Cypher Investigators. Safety of coronary sirolimus-eluting stents in daily clinical practice: one-year follow-up of the e-Cypher registry. Circulation. 2006 Mar 21;113(11):1434-41. doi: 10.1161/CIRCULATIONAHA.104.532242. Epub 2006 Mar 13. PMID 16534015
- [Background] Schampaert E, Cohen EA, Schluter M, Reeves F, Traboulsi M, Title LM, Kuntz RE, Popma JJ; C-SIRIUS Investigators. The Canadian study of the sirolimus-eluting stent in the treatment of patients with long de novo lesions in small native coronary arteries (C-SIRIUS). J Am Coll Cardiol. 2004 Mar 17;43(6):1110-5. doi: 10.1016/j.jacc.2004.01.024. PMID 15028375
- [Background] Lemos PA, Serruys PW, van Domburg RT, Saia F, Arampatzis CA, Hoye A, Degertekin M, Tanabe K, Daemen J, Liu TK, McFadden E, Sianos G, Hofma SH, Smits PC, van der Giessen WJ, de Feyter PJ. Unrestricted utilization of sirolimus-eluting stents compared with conventional bare stent implantation in the "real world": the Rapamycin-Eluting Stent Evaluated At Rotterdam Cardiology Hospital (RESEARCH) registry. Circulation. 2004 Jan 20;109(2):190-5. doi: 10.1161/01.CIR.0000109138.84579.FA. Epub 2003 Dec 22. PMID 14691037
- [Background] Daemen J, Serruys PW. Drug-eluting stent update 2007: part I. A survey of current and future generation drug-eluting stents: meaningful advances or more of the same? Circulation. 2007 Jul 17;116(3):316-28. doi: 10.1161/CIRCULATIONAHA.106.621342. No abstract available. PMID 17638940
- [Background] Sousa JE, Costa MA, Abizaid A, Abizaid AS, Feres F, Pinto IM, Seixas AC, Staico R, Mattos LA, Sousa AG, Falotico R, Jaeger J, Popma JJ, Serruys PW. Lack of neointimal proliferation after implantation of sirolimus-coated stents in human coronary arteries: a quantitative coronary angiography and three-dimensional intravascular ultrasound study. Circulation. 2001 Jan 16;103(2):192-5. doi: 10.1161/01.cir.103.2.192. PMID 11208675
- [Background] Poon M, Marx SO, Gallo R, Badimon JJ, Taubman MB, Marks AR. Rapamycin inhibits vascular smooth muscle cell migration. J Clin Invest. 1996 Nov 15;98(10):2277-83. doi: 10.1172/JCI119038. PMID 8941644
- [Background] Moses JW, Leon MB, Popma JJ, Fitzgerald PJ, Holmes DR, O'Shaughnessy C, Caputo RP, Kereiakes DJ, Williams DO, Teirstein PS, Jaeger JL, Kuntz RE; SIRIUS Investigators. Sirolimus-eluting stents versus standard stents in patients with stenosis in a native coronary artery. N Engl J Med. 2003 Oct 2;349(14):1315-23. doi: 10.1056/NEJMoa035071. PMID 14523139
- [Background] Morice MC, Serruys PW, Barragan P, Bode C, Van Es GA, Stoll HP, Snead D, Mauri L, Cutlip DE, Sousa E. Long-term clinical outcomes with sirolimus-eluting coronary stents: five-year results of the RAVEL trial. J Am Coll Cardiol. 2007 Oct 2;50(14):1299-304. doi: 10.1016/j.jacc.2007.06.029. Epub 2007 Sep 17. PMID 17903626
- [Background] Klugherz BD, Llanos G, Lieuallen W, Kopia GA, Papandreou G, Narayan P, Sasseen B, Adelman SJ, Falotico R, Wilensky RL. Twenty-eight-day efficacy and phamacokinetics of the sirolimus-eluting stent. Coron Artery Dis. 2002 May;13(3):183-8. doi: 10.1097/00019501-200205000-00008. PMID 12131023
- [Background] Sousa JE, Costa MA, Abizaid A, Feres F, Seixas AC, Tanajura LF, Mattos LA, Falotico R, Jaeger J, Popma JJ, Serruys PW, Sousa AG. Four-year angiographic and intravascular ultrasound follow-up of patients treated with sirolimus-eluting stents. Circulation. 2005 May 10;111(18):2326-9. doi: 10.1161/01.CIR.0000164271.01172.1A. Epub 2005 Apr 25. PMID 15851603
- [Background] Popma JJ, Topol EJ. Factors influencing restenosis after coronary angioplasty. Am J Med. 1990 Jan;88(1N):16N-24N. PMID 2195881
- [Background] Stone GW, Ellis SG, Colombo A, Dawkins KD, Grube E, Cutlip DE, Friedman M, Baim DS, Koglin J. Offsetting impact of thrombosis and restenosis on the occurrence of death and myocardial infarction after paclitaxel-eluting and bare metal stent implantation. Circulation. 2007 Jun 5;115(22):2842-7. doi: 10.1161/CIRCULATIONAHA.106.687186. Epub 2007 May 21. PMID 17515458
- [Background] Kastrati A, Mehilli J, Dirschinger J, Pache J, Ulm K, Schuhlen H, Seyfarth M, Schmitt C, Blasini R, Neumann FJ, Schomig A. Restenosis after coronary placement of various stent types. Am J Cardiol. 2001 Jan 1;87(1):34-9. doi: 10.1016/s0002-9149(00)01268-6. PMID 11137830
- [Background] Doostzadeh J, Clark LN, Bezenek S, Pierson W, Sood PR, Sudhir K. Recent progress in percutaneous coronary intervention: evolution of the drug-eluting stents, focus on the XIENCE V drug-eluting stent. Coron Artery Dis. 2010 Jan;21(1):46-56. doi: 10.1097/MCA.0b013e328333f550. PMID 19952925
- [Background] Serruys PW, Regar E, Carter AJ. Rapamycin eluting stent: the onset of a new era in interventional cardiology. Heart. 2002 Apr;87(4):305-7. doi: 10.1136/heart.87.4.305. No abstract available. PMID 11906992
- [Background] Suzuki T, Kopia G, Hayashi S, Bailey LR, Llanos G, Wilensky R, Klugherz BD, Papandreou G, Narayan P, Leon MB, Yeung AC, Tio F, Tsao PS, Falotico R, Carter AJ. Stent-based delivery of sirolimus reduces neointimal formation in a porcine coronary model. Circulation. 2001 Sep 4;104(10):1188-93. doi: 10.1161/hc3601.093987. PMID 11535578
- [Background] Sousa JE, Costa MA, Farb A, Abizaid A, Sousa A, Seixas AC, da Silva LM, Feres F, Pinto I, Mattos LA, Virmani R. Images in cardiovascular medicine. Vascular healing 4 years after the implantation of sirolimus-eluting stent in humans: a histopathological examination. Circulation. 2004 Jul 6;110(1):e5-6. doi: 10.1161/01.CIR.0000134307.00204.B3. No abstract available. PMID 15238468